CLINICAL TRIAL: NCT07103811
Title: The Relationship Between Social Media Use, Food Craving and Ultra-Processed Food Consumption in University Students
Brief Title: Social Media Use, Food Craving and Ultra Processed Food Consumption in Students
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: Sedef Güngör-Atılım-03
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Food Craving; Ultra Processed Food; Social Media
Keywords: Food craving; Ultra processed food; Social media

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Social media can increase unhealthy eating habits by influencing individuals' desire to eat, especially through images and advertisements of ultra-processed foods. One of the groups most affected by this situation is university students who use social media intensively. Therefore, examining the relationship between social media use and ultra-processed food consumption is important in terms of developing healthy eating awareness.

DETAILED DESCRIPTION:
Nowadays, social media has gained an important place in the daily lives of individuals and has become a factor that can be effective on dietary habits. Food content frequently shared on social media platforms, especially advertisements related to ultra-processed foods, can shape food perceptions and consumption behaviours. This may increase ultra-processed food consumption by triggering individuals' food craving.

Ultra-processed foods are foods that contain high levels of sugar, fat, salt and additives, have low nutritional value but are attractive in terms of flavour. Such foods can create an addiction-like consumption cycle because they provide fast energy and directly affect the brain reward system. Intensive visual and content exposure to these foods on social media may increase individuals' appetite reactions and lead to the spread of unhealthy eating habits.

University students are one of the most affected groups due to their young age group and intensive use of social media. At the same time, it is known that the eating habits acquired during this period are decisive on sustainable health in the long term. Therefore, examining the relationship between social media use, food craving and ultra-processed food consumption is an important issue in terms of developing nutritional awareness and promoting healthy eating habits.

Objective: This study aims to examine the effect of university students' exposure to ultra-processed food content on their food craving and ultra-processed food consumption on social media platforms.

Method This study will be conducted online via a questionnaire prepared through Google Forms and the students of Atılım University will be included in the study. Before starting the study, participants will be asked to read and approve the Informed Voluntary Consent Form. The study will be conducted with at least 150 participants. It is planned to collect and analyse the data between April 2025 and June 2025.

The first part of the data collection form includes questions about the demographic characteristics (gender, age, marital status, occupation, etc.) and anthropometric measurements (body weight, height) of the participants. In the second part of the form, there will be questions about their social media use (duration of use, exposure to nutrients, etc.). The third part of the questionnaire form includes the 'Food Craving Questionnaire Short Form (FCQT-R)', which was developed to evaluate the desire to eat and was adapted into Turkish in 2021. The scale consists of 15 questions and includes a 6-point scale ranging from 'Never' (1) to 'Always' (6). The scale has a score range of 15-90. A low score indicates a low food craving experience, while a high score indicates a high food craving experience. In the fourth part of the data collection form, the 'Multiprocessed Food Consumption Short Screening Questionnaire' developed for the evaluation of ultra-processed food consumption and adapted into Turkish by Gövez et al. There are 11 items in the scale. For each question, the participants will be asked to tick one of the yes or no answers. The score that can be obtained from the scale varies between 0 and 11. There are no reverse items in the scale. Each yes is scored as 1 point. 6 points and above is considered as high processed food consumption. Participants will not be asked for their names and identity information, and research data will not be shared with any institution.

Expected Results of the Study: This study is expected to show that exposure to ultra-processed food content on social media may increase university students' food craving and ultra-processed food consumption. It is predicted that the duration of social media use and content interaction may encourage unconscious eating behaviours and this may lead to unhealthy eating habits. The findings are expected to contribute to understanding the effects of social media on nutrition and shed light on the development of strategies that promote healthy eating.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-25
* To reside in Ankara
* Being a university student
* Volunteering
* No communication problems

Exclusion Criteria:

* Under 18 years of age and over 25 years of age
* Persons who are not university students
* Those who do not reside in Ankara
* Those with communication problems
* Having any psychological disorder

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: The population of this study consisted of male and female university students aged between 18 and 25 years studying in Ankara.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the correlation between social media use and ultra-processed food consumption in university students | Up to one month
  Questions about students' social media use (duration of use, exposure to nutrients, etc.) will be collected with a questionnaire form. In order to evaluate ultra-processed food consumption, 'short screening questionnaire of highly processed food consumption (sQ-HPF)' will be applied. There are 11 items in the scale. For each question, the participants will be asked to tick one of the yes or no answers. The score that can be obtained from the scale varies between 0 and 11. There is no reverse item in the scale. Each yes is evaluated as 1 point. 6 points and above is considered as high processed food consumption.
Evaluation of the correlation between Social Media Use and Food Craving in University Students | Up to one month
  Questions about students' social media use (duration of use, exposure to foods, etc.) will be collected with a questionnaire form. 'Food Craving Questionnaire Short Form (FCQT-R)' will be used to evaluate the desire to eat. The scale consists of 15 questions and includes a 6-point scale ranging from "Never" (1) to "Always" (6). The scale has a score range of 15-90. A low score indicates a low food craving experience, while a high score indicates a high food craving experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Aleid S, Alshahrani NZ, Alsedrah S, Carvalho AB, Lima MJ, Teixeira-Lemos E, Raposo A. The Role of Social Media Advertisement and Physical Activity on Eating Behaviors among the General Population in Saudi Arabia. Nutrients. 2024 Apr 19;16(8):1215. doi: 10.3390/nu16081215. PMID 38674905
- [Background] Filippone L, Shankland R, Hallez Q. The relationships between social media exposure, food craving, cognitive impulsivity and cognitive restraint. J Eat Disord. 2022 Nov 25;10(1):184. doi: 10.1186/s40337-022-00698-4. PMID 36434703
- [Background] Cheikh Ismail L, Osaili TM, Naja F, Wartanian M, Elkabat G, Arnous M, Alkoukou H, Mohamad MN, Saleh ST, Al Daour R, Masuadi E, Ali HI, Stojanovska L, Al Dhaheri AS. The association of social media with dietary behaviors among adults in the United Arab Emirates. Heliyon. 2024 Jul 31;10(15):e35574. doi: 10.1016/j.heliyon.2024.e35574. eCollection 2024 Aug 15. PMID 39166066
- [Background] Fondevila-Gascon JF, Berbel-Gimenez G, Vidal-Portes E, Hurtado-Galarza K. Ultra-Processed Foods in University Students: Implementing Nutri-Score to Make Healthy Choices. Healthcare (Basel). 2022 May 25;10(6):984. doi: 10.3390/healthcare10060984. PMID 35742036
- [Background] Cepeda-Benito A, Gleaves DH, Fernandez MC, Vila J, Williams TL, Reynoso J. The development and validation of Spanish versions of the State and Trait Food Cravings Questionnaires. Behav Res Ther. 2000 Nov;38(11):1125-38. doi: 10.1016/s0005-7967(99)00141-2. PMID 11060941
- [Background] Meule A, Hermann T, Kubler A. A short version of the Food Cravings Questionnaire-Trait: the FCQ-T-reduced. Front Psychol. 2014 Mar 4;5:190. doi: 10.3389/fpsyg.2014.00190. eCollection 2014. PMID 24624116
- [Background] Martinez-Perez C, Daimiel L, Climent-Mainar C, Martinez-Gonzalez MA, Salas-Salvado J, Corella D, Schroder H, Martinez JA, Alonso-Gomez AM, Warnberg J, Vioque J, Romaguera D, Lopez-Miranda J, Estruch R, Tinahones FJ, Lapetra J, Serra-Majem L, Bueno-Cavanillas A, Tur JA, Sanchez VM, Pinto X, Delgado-Rodriguez M, Matia-Martin P, Vidal J, Vazquez C, Ros E, Basterra J, Babio N, Guillem-Saiz P, Zomeno MD, Abete I, Vaquero-Luna J, Baron-Lopez FJ, Gonzalez-Palacios S, Konieczna J, Garcia-Rios A, Bernal-Lopez MR, Santos-Lozano JM, Bes-Rastrollo M, Khoury N, Saiz C, Perez-Vega KA, Zulet MA, Tojal-Sierra L, Ruiz ZV, Martinez MA, Malcampo M, Ordovas JM, San-Cristobal R. Integrative development of a short screening questionnaire of highly processed food consumption (sQ-HPF). Int J Behav Nutr Phys Act. 2022 Jan 24;19(1):6. doi: 10.1186/s12966-021-01240-6. PMID 35073909
- [Background] Erdogan Govez N, Koksal E, Martinez-Perez C, Daimiel L. Validity and Reliability of the Turkish Version of the Screening Questionnaire of Highly Processed Food Consumption (sQ-HPF). Nutrients. 2024 Aug 3;16(15):2552. doi: 10.3390/nu16152552. PMID 39125430